CLINICAL TRIAL: NCT06213974
Title: Post Authorization Study to Monitor Efficacy, Effectiveness, and Safety of Maribavir (LIVTENCITY®) in Patients With Post-transplant Cytomegalovirus (CMV) Infection in Argentina
Brief Title: A Study of Maribavir in Adults and Children With Post-transplant Cytomegalovirus (CMV) Infection in Argentina
Status: Recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-620-4008
Record Dates: First submitted 2024-01-10; First posted 2024-01-19 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Cytomegalovirus (CMV)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: Participants who have received maribavir treatment for the approved indication after marketing authorization (de novo participants) and before marketing authorization (legacy participants) under expanded access type of program or compassionate use in the real-world setting. Data will be collected prospectively and/or retrospectively from the medical records during this observational period of 16 weeks.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is non-interventional study.

SUMMARY:
The main aim of this study is to learn about the safety of Maribavir in adults and children with post-transplant CMV infection in routine clinical practice in Argentina.

The other aim is to study the effectiveness of the treatment with Maribavir in routine clinical practice in Argentina.

Participants will be treated by their doctors according to normal medical practice. Study data will be collected either from information already available in the medical records or during study conduct.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (18 years or older) and pediatric participants (12 years of age and older and weighing at least 35 kilogram [kg]) with post-transplant CMV infection/disease that is refractory to treatment (with or without genotypic resistance) with ganciclovir, valganciclovir, cidofovir or foscarnet in the real-world setting of common clinical practice in Argentina.
* Have received at least one dose of maribavir according to approved indications.
* Have signed the mandatory informed consent/assent that has been agreed with national regulatory authorities (ANMAT) as applicable.

Exclusion Criteria

- There are no specific exclusion criteria.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and pediatric participants with post-transplant CMV infection/disease that are refractory to treatment (with or without genotypic resistance) with ganciclovir, valganciclovir, cidofovir or foscarnet, that are treated with maribavir according to approved indications.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | From start of treatment up to Week 16
  An AE is any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which does not necessarily have a causal relationship with this treatment. AEs will include both serious and non-serious AEs.

SECONDARY OUTCOMES:
Percentage of Participants Who Achieved Clearance of Plasma Cytomegalovirus -Deoxyribonucleic Acid (CMV-DNA) (CMV Viremia Clearance) at End of Weeks 8 and 16 | At Weeks 8 and 16
  CMV viremia clearance will be defined as CMV DNA concentration below the lower limit of considered by each local site for clearance according to real-world clinical practice.
Percentage of Participants Who Achieved CMV Infection Symptom Control at End of Weeks 8 and 16 | At Weeks 8 and 16
  CMV infection symptom control will be defined as resolution or improvement CMV disease/syndrome for participants symptomatic at baseline, or absence of the development of CMV disease/syndrome or participants asymptomatic at baseline.
Percentage of Participants Who Achieved a Clinically Relevant Response Regardless of Whether Treatment was Discontinued Before 8 weeks of Therapy | Up to Week 8
  Clinically relevant response will be defined as no need for the use of an antiviral at a therapeutic dose for at least 4 weeks after completing treatment with maribavir, due to clinical improvement (improvement of CMV-related symptoms or the absence of these in the case of asymptomatic infections) and virological improvement (decrease of at least 1 log of viremia during treatment with maribavir).

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (1):
- IC Projects, City of Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click this link. — https://clinicaltrials.takeda.com/study-detail/761e35a0e7fa48a0??page=1&idFilter=TAK-620-4008